CLINICAL TRIAL: NCT00666614
Title: A Pilot Study to Examine Sleep and Fatigue in Pediatric Brain Tumor Patients Hospitalized for High Dose Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BTSLEP
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2012-01

CONDITIONS: Sleep; Fatigue
Keywords: Sleep; Fatigue; High Dose Chemotherapy
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): Patients randomized to the sleep environment intervention months will experience a relaxation period before nighttime sleep, white noise as selected by the patient, stimulus control strategies, a window covering to diminish hallway light from entering the room, and a nurse-protected 90-minute uninterrupted sleep period at night.
  Interventions: Other: Sleep Environment Intervention
- Standard Care (Other): Normal Hospital Environment
  Interventions: Other: Normal Hospital Environment

INTERVENTIONS:
Other: Sleep Environment Intervention — Patients randomized to the sleep environment intervention months will experience a relaxation period before nighttime sleep, white noise as selected by the patient, stimulus control strategies, a window covering to diminish hallway light from entering the room, and a nurse-protected 90-minute uninterrupted sleep period at night.
  Arms: Intervention
Other: Normal Hospital Environment — Normal Hospital Environment
  Arms: Standard Care

SUMMARY:
The purpose of this pilot study is to determine if patients randomized to a hospital sleep environment intervention would have improved sleep quality and reduced fatigue as compared to the patients not receiving the intervention (standard care).

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if patients randomized to a hospital sleep environment intervention would have improved sleep quality and reduced fatigue as compared to the patients not receiving the intervention (standard care).

All patients enrolled on SJMB03 and admitted to receive either the 2nd or 3rd course of chemotherapy will be eligible for the study. The patients are admitted for four to six days and all participants will wear an actigraph to collect information on 8 sleep quality indicators for each of the six days. In addition, fatigue measurements will also be collected and compared between the two groups. Given the nature of the intervention, it is difficult to follow the traditional randomization scheme and randomize eligible patients to the intervention or standard care because there is a high likelihood of design contamination secondary to interactions among family members and among the nurses in regards to the different care for the study participants in the two study groups. Therefore, this study will use a group randomized trial design with patients randomized by month. That is, all patients admitted in a month randomized to be an intervention month will receive the intervention and all patients admitted to a standard care month will not receive the intervention. This type of randomization plan has notable strengths that match this study design but it also has two potential challenges: 1) patients randomized within the last five days of each month will continue to receive the assigned treatment to which they were randomized although this treatment assignment will continue into a different month that could have been randomized to the same or different condition as the previous month, and 2) with random assignments of months to the two treatment arms, there is a possibility of an unequal distribution of patients randomized to the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 4 and 21 years who are enrolled on SJMB03 and to be admitted for either Course 2 or Course 3 of high dose chemotherapy and stem cell rescue.
* English - speaking and able to understand English items on the study instruments as these are only available in English.
* Patients willing to give assent to participate in the study and whose parents are willing to give permission according to institutional guidelines for their child to participate.

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Patients experiencing serious neurological effects such as posterior fossa syndrome that interfere with their ability to self-report on fatigue and mood.
* Patient is bedridden and unable to participate in an activity.
* Patients or parents who would find participating in the consent process too emotionally demanding as determined by the treatment team.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess sleep quality, fatigue and daytime activity during the 4 to 6-day hospitalization as being more positive for patients randomized to the sleep environment intervention months as compared to those randomized to the standard care months | Within 6 -10 months

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Mandrell, PhD, RN, PNP, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] Graef DM, Crabtree VM, Srivastava DK, Li C, Pritchard M, Hinds PS, Mandrell B. Sleep and mood during hospitalization for high-dose chemotherapy and hematopoietic rescue in pediatric medulloblastoma. Psychooncology. 2018 Jul;27(7):1847-1853. doi: 10.1002/pon.4737. Epub 2018 May 16. PMID 29663636
- [Result] Rogers VE, Zhu S, Mandrell BN, Ancoli-Israel S, Liu L, Hinds PS. Relationship between circadian activity rhythms and fatigue in hospitalized children with CNS cancers receiving high-dose chemotherapy. Support Care Cancer. 2020 Mar;28(3):1459-1467. doi: 10.1007/s00520-019-04960-5. Epub 2019 Jul 4. PMID 31273507
- [Result] Rogers VE, Zhu S, Ancoli-Israel S, Liu L, Mandrell BN, Hinds PS. A pilot randomized controlled trial to improve sleep and fatigue in children with central nervous system tumors hospitalized for high-dose chemotherapy. Pediatr Blood Cancer. 2019 Aug;66(8):e27814. doi: 10.1002/pbc.27814. Epub 2019 May 13. PMID 31081596
- See also: St. Jude Children's Research Hospital — http://www.stjude.org